CLINICAL TRIAL: NCT04858997
Title: An Open-label, Prospective Study of Tumor Response Time of Palbociclib in Combination With AI in Real-world First-line Treatment of Postmenopausal Chinese Patients With ER (+) HER2 (-) Metastatic Breast Cancer
Brief Title: Tumor Response Time of Palbociclib in Combination With AI in Real-world Chinese Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-ZJCC-02
Record Dates: First submitted 2021-03-24; First posted 2021-04-26 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib-AI (Experimental): ER(+)/HER2(-) patients with histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease receive palbociclib PO daily on days 1-21, combined with AI as first-line treatment Disease assessments measured by CT imaging will be performed at first 4 weeks, 8weeks, then every 8weeks (± 7 days) from the date of randomization until radiographic/clinical documentation of progressive disease per the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
  Interventions: Drug: Palbociclib; Drug: AI

INTERVENTIONS:
Drug: Palbociclib — Palbociclib,125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Other Names: Ibrabce
Drug: AI — AI, orally once daily (continuously)

SUMMARY:
The international treatment guidelines now include recommendations for the use of CDK 4/6 inhibitors in combination with hormone agents for the treatment of postmenopausal women with hormone-receptor-positive/HER2-negative ABC as the first-line standard therapy in endocrine sensitive patients.

Nevertheless, it is generally thought that chemotherapy is associated with greater and earlier tumor response, especially in case of high burden of disease. In a retrospective analysis of real-world clinical practice (2002-2012) from US, only 60% of patients initiated ET as the first treatment following metastatic diagnosis . In the real-life world of China, a large number of HR+/HER2- ABC patients with non-visceral crisis also received chemotherapy in first-line treatment, even though the ORR is similar compared with CDK4/6 inhibitors with endocrine therapy. Zhejiang Cancer Hospital retrospective analysis of 5 cases of advanced breast cancer first-line use of Ibance + ET, they were evaluated within 50 days (from 27days to 50days).

Based on the early response time observed in real-world data mentioned above, it is proposed a prospective study to further observe the tumor reduction rate in real-world, including to identify the time of patient symptom improvement according to the quality of life scale.

DETAILED DESCRIPTION:
According to the early assessment(4 weeks) , this prospective study comprehensively investigate TTR of Palbociclib+ET in the first line treatment for HR+/HER2- MBC patients in China real-world study.

Furthermore, evaluate the Early Tumor Shrinkage(ETS) of Palbociclib + ET, and assess Treatment Free Interval (TFI) with TTR and ETS；TFI was analyzed at the following time points: ≤24, >24, ≤36, > 36, ≤48, >48 months.

Accroding to the follow-up of QoL questionnaire, understand the clinical symptoms improvements time.

Meanwhile, cooperation with radiology department, establish a model for predicting early response by observing the imaging and clinical pathological characteristics of patients with ETS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 18 years of age) with proven diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent and for whom chemotherapy is not clinically indicated.
2. Documentation of histologically or cytologically confirmed diagnosis of estrogen-receptor positive (ER+, > 10%) breast cancer based on local laboratory results.
3. Previously untreated with any systemic anti-cancer therapy for their locoregionally recurrent or metastatic ER+ disease.
4. Postmenopausal women.
5. At least one measurable lesion as defined per RECIST v.1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
7. Adequate organ and marrow function.
8. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with advanced, symptomatic, visceral spread, that are at risk of life-threatening complications including any of the following:

   * massive uncontrolled effusions [pleural, pericardial, peritoneal]
   * pulmonary lymphangitis,
   * over 50% liver involvement
2. Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis,or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.
3. Prior neoadjuvant or adjuvant treatment with a non-steroidal aromatase inhibitor (ie, anastrozole or letrozole) with disease recurrence while on or within 12 months of completing treatment.
4. Prior treatment with any CDK4/6 inhibitor.
5. QTc >480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
6. Female patients who are pregnant or nursing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal
Enrollment: 150 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Early Tumor Shrinkage (ETS) | 4 weeks, 8weeks
  10% change in the sum of the longest diameters (SLD) of target lesions at the first scan after 4weeks and 8weeks of treatment.
Time To Response (TTR) | Up to approximately 24 months
  Time to first documented complete of partial response.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the overall complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1)
Number of participants with Adverse Events per CTCAE version 4.03 and type | Up to approximately 24 months
  Safety will be determined by type, severity of adverse events per CTCAE version 4.03 and type
Time to Definitive 10% Deterioration in the Global Health Status/Quality of Life (QOL) Scale Score of the EORTC QLQ-C30 | Up to approximately 24 months
  At least 10% relative to baseline worsening of the corresponding scale score (without further improvement above the threshold) or death due to any cause.
Overall Survival (OS) | Randomization to death from any cause, through the end of study (approximately 60months)]
  time to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ming Cao, Ph.D., M.D., Principal Investigator — Department of Breast Medical Oncology, Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lobbezoo DJ, van Kampen RJ, Voogd AC, Dercksen MW, van den Berkmortel F, Smilde TJ, van de Wouw AJ, Peters FP, van Riel JM, Peters NA, de Boer M, Borm GF, Tjan-Heijnen VC. Prognosis of metastatic breast cancer subtypes: the hormone receptor/HER2-positive subtype is associated with the most favorable outcome. Breast Cancer Res Treat. 2013 Oct;141(3):507-14. doi: 10.1007/s10549-013-2711-y. Epub 2013 Oct 9. PMID 24104881
- [Result] Cardoso F, Senkus E, Costa A, Papadopoulos E, Aapro M, Andre F, Harbeck N, Aguilar Lopez B, Barrios CH, Bergh J, Biganzoli L, Boers-Doets CB, Cardoso MJ, Carey LA, Cortes J, Curigliano G, Dieras V, El Saghir NS, Eniu A, Fallowfield L, Francis PA, Gelmon K, Johnston SRD, Kaufman B, Koppikar S, Krop IE, Mayer M, Nakigudde G, Offersen BV, Ohno S, Pagani O, Paluch-Shimon S, Penault-Llorca F, Prat A, Rugo HS, Sledge GW, Spence D, Thomssen C, Vorobiof DA, Xu B, Norton L, Winer EP. 4th ESO-ESMO International Consensus Guidelines for Advanced Breast Cancer (ABC 4)dagger. Ann Oncol. 2018 Aug 1;29(8):1634-1657. doi: 10.1093/annonc/mdy192. No abstract available. PMID 30032243
- [Result] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Result] Swallow E, Zhang J, Thomason D, Tan RD, Kageleiry A, Signorovitch J. Real-world patterns of endocrine therapy for metastatic hormone-receptor-positive (HR+)/human epidermal growth factor receptor-2-negative (HER2-) breast cancer patients in the United States: 2002-2012. Curr Med Res Opin. 2014 Aug;30(8):1537-45. doi: 10.1185/03007995.2014.908829. Epub 2014 Apr 14. PMID 24669852
- [Result] Turner NC, Finn RS, Martin M, Im SA, DeMichele A, Ettl J, Dieras V, Moulder S, Lipatov O, Colleoni M, Cristofanilli M, Lu DR, Mori A, Giorgetti C, Iyer S, Bartlett CH, Gelmon KA. Clinical considerations of the role of palbociclib in the management of advanced breast cancer patients with and without visceral metastases. Ann Oncol. 2018 Mar 1;29(3):669-680. doi: 10.1093/annonc/mdx797. PMID 29342248
- [Result] Piessevaux H, Buyse M, Schlichting M, Van Cutsem E, Bokemeyer C, Heeger S, Tejpar S. Use of early tumor shrinkage to predict long-term outcome in metastatic colorectal cancer treated with cetuximab. J Clin Oncol. 2013 Oct 20;31(30):3764-75. doi: 10.1200/JCO.2012.42.8532. Epub 2013 Sep 16. PMID 24043732
- [Result] Wei M, Ye Q, Wang X, Wang M, Hu Y, Yang Y, Yang J, Cai J. Early tumor shrinkage served as a prognostic factor for patients with stage III non-small cell lung cancer treated with concurrent chemoradiotherapy. Medicine (Baltimore). 2018 May;97(19):e0632. doi: 10.1097/MD.0000000000010632. PMID 29742701
- [Result] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Result] Janni W, Alba E, Bachelot T, Diab S, Gil-Gil M, Beck TJ, Ryvo L, Lopez R, Tsai M, Esteva FJ, Aunon PZ, Kral Z, Ward P, Richards P, Pluard TJ, Sutradhar S, Miller M, Campone M. First-line ribociclib plus letrozole in postmenopausal women with HR+ , HER2- advanced breast cancer: Tumor response and pain reduction in the phase 3 MONALEESA-2 trial. Breast Cancer Res Treat. 2018 Jun;169(3):469-479. doi: 10.1007/s10549-017-4658-x. Epub 2018 Feb 5. PMID 29404806